CLINICAL TRIAL: NCT05661617
Title: The Influence of Laterality on the Performance of Healthy Women Aged 20-24 Years in Selected Standardized Tests Assessing the Upper Limbs Function
Brief Title: The Influence of Laterality on the Performance of Healthy Women in Selected Standardized Tests
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, occupational therapist, lecturer, Charles University, Czech Republic
Other Study IDs: 219/22 S-IV
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Motor Activity
Keywords: fine motor skills; occupational therapy; Nine Hole Peg Test; Purdue Pegboard Test; Box and Block Test
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Czech healthy women tested in normative study: Czech healthy women aged 20-24 years tested in study called "Establishing Czech Norms of Selected Standardized Tests".
  Interventions: Diagnostic Test: Nine Hole Peg Test, Purdue Pegboard Test, Box and Block Test
- Czech healthy women (experimental group): Czech healthy women aged 20-24 years (inclusive) who participated in the research in the period from January 2023.
  Interventions: Diagnostic Test: Nine Hole Peg Test, Purdue Pegboard Test, Box and Block Test

INTERVENTIONS:
Diagnostic Test: Nine Hole Peg Test, Purdue Pegboard Test, Box and Block Test — Research participants were tested in one meeting after giving informed consent, answering a few short questions regarding health status and filling out a short questionnaire using the Czech extended version of the manual for the Nine Hole Peg Test, Purdue Pegboard Test and Box and Block Test, and always according to a predetermined order. Intentionally, all research participants from experimental group with a dominant right upper limb will be tested as if they were left-handed, and vice versa.
  All research participants from normative study were tested normally according to the Czech extended manuals for those tests.

SUMMARY:
The aim of the research study is to find out how the results of healthy women aged 20-24 years (inclusive) differ in the Nine Peg Test, the Purdue Pegboard Test and the Box and Block Test, depending on the laterality of the research participants and the order of the performed subtests of the investigated tests. In this way, it will be preliminarily determined whether it is necessary to create normative data separately for right-handed and left-handed people for the tests.

DETAILED DESCRIPTION:
Research participants will be tested in one meeting after giving informed consent, answering a few short questions regarding health status and filling out a short questionnaire using the Czech extended version of the manual for all three standardized tests, and always according to a predetermined order. Intentionally, all research participants with a dominant right upper limb will be tested as if they were left-handed, and vice versa.

The results of the research participants tested in this way will be compared with the results of women from the same age category who have already been properly tested as part of an ongoing research study entitled: "Establishing Czech Norms of Selected Standardized Tests".

ELIGIBILITY:
Inclusion Criteria:

* Czech language as a mother tongue
* age from 20 to 24 years (inclusive)
* female

Exclusion Criteria:

* diagnosed pathology of the upper limbs or diseases that negatively affect the dexterity of their limbs
* use of drugs affecting attention
* vision impairment uncorrectable with glasses
* severe hearing loss
* inability to understand instructions
* inability to read or write
* inability to complete testing
* failure to sign Informed consent for probation with inclusion to research and Consent to the collection and processing of personal data during the study at the General University Hospital in Prague

Ages: 20 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: healthy women from the Czech Republic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
results from the Nine Hole Peg Test | 10 minutes
  time in seconds and hundreds of seconds
results from the Purdue Pegboard Test | 25 minutes
  number of parts put in the Pegboard according to the rules
results from the Box and Block Test | 30 minutes
  number of transported blocks

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Rybářová, Mgr., Study Director — Charles University, Czech Republic
Locations (1):
- Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No